CLINICAL TRIAL: NCT00024102
Title: A Randomized Trial of Adjuvant Chemotherapy With Standard Regimens, Cyclophosphamide, Methotrexate and Fluorouracil - (CMF) or Doxorubicin and Cyclophosphamide - (AC), Versus Capecitabine in Women 65 Years and Older With Node Positive or Node-Negative Breast Cancer
Brief Title: Comparison of Combination Chemotherapy Regimens in Treating Older Women Who Have Undergone Surgery for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-49907; U10CA031946 (NIH); CAN-NCIC-MAC1; CDR0000068891 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Chemotherapy (Active Comparator): Patient/Physician choice of cyclophosphamide + MTX + 5-FU
  OR
  Cyclophosphamide + doxorubicin
  Interventions: Drug: Standard Treatment
- Capecitabine (Experimental): Treatment with capecitabine
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Standard Treatment — Cyclophosphamide 100 mg/sq m PO d 1-14 + MTX 40 mg/sq m IV push d 1 & 8 and 5-FU 600 mg/sq m IV push d 1 & 8 q 28 days for 6 cycles OR doxorubicin 60 mg/sq m IV d 1 + cyclophosphamide 600 mg/sq m IV d 1 q 21 d for 4 cycles
  Other Names: doxorubicin = adriamycin
  Arms: Standard Chemotherapy
Drug: capecitabine — 2000 mg/sq m PO d 1-14, 7 day rest then repeat for a total of 6 cycles
  Arms: Capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways after surgery may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective in treating older women with breast cancer.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens to see how well they work in treating older women who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of adjuvant chemotherapy comprising standard cyclophosphamide, methotrexate, and fluorouracil (CMF) or doxorubicin and cyclophosphamide (AC) vs oral capecitabine, in terms of disease-free and overall survival, in elderly women with operable adenocarcinoma of the breast.
* Compare the quality of life and physical functioning of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Evaluate the adherence of older patients to an oral chemotherapy regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (65 to 69 vs 70 to 80 vs over 80), performance status (0-1 vs 2), and HER2 status (positive vs negative vs unknown). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients with insufficient left ventricular ejection fraction (LVEF) are assigned to group A. Patients with normal LVEF are assigned to group A or B based on physician/patient choice.

  * Group A (CMF): Patients receive oral cyclophosphamide (CTX) daily on days 1-14 and methotrexate IV and fluorouracil IV on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Group B (AC): Patients receive doxorubicin IV and CTX IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Beginning within 12 weeks after treatment in arm I or II, patients with estrogen or progesterone receptor-positive disease receive oral tamoxifen or an aromatase inhibitor daily for 5 years.

Beginning 4-6 weeks after treatment in arm I or II, eligible patients who previously underwent breast conservation surgery undergo radiotherapy.

Quality of life is assessed at baseline; at 6 weeks (group B), 9 weeks (arm II), or 12 weeks (group A); and then at 1, 12, 18, and 24 months after study.

Drug adherence is assessed at 9 weeks during study (arm II).

Patients are followed at 1 month, every 6 months for 2 years, and then annually for 15 years.

PROJECTED ACCRUAL: A total of 600-1,800 patients (300-900 per treatment arm) will be accrued for this study within 2-6 years.

ELIGIBILITY:
1. Patients with operable, histologically confirmed adenocarcinoma of the female breast.
2. TNM Stage per AJCC Cancer Staging Manual 6th edition:

   * T1-4 (Tumor size > 1 cm), N0, M0 or T1-4, N1-3, M0
   * Patients with bilateral, synchronous breast cancer are eligible as long as one primary tumor meets the criteria above.
3. Patients with HER2/neu positive, negative or unknown disease are eligible for this trial.

   Patients whose tumors are HER2 positive by either immunohistochemistry 3+ staining or demonstrate gene amplification by FISH will be eligible to receive trastuzumab, as outlined in the protocol.
4. Age 65 years or older
5. Performance status 0-2 (Common Toxicity Criteria).
6. Prior treatment:

   * Surgical resection -

     * All tumor should be removed by either a modified radical mastectomy or a lumpectomy. Patients must be registered ≤ 84 days from mastectomy or within 84 days of axillary dissection if patient's most extensive breast surgery was a breast sparing procedure.
     * Node dissection: Axillary node dissection is not required. Management of the axilla is at the discretion of the treating physician. There is no restriction on eligibility based on the number of nodes removed.
     * Mastectomy: There should be no evidence of gross or microscopic invasive tumor at the surgical resection margins noted in the final surgery or pathology reports for patients who have had a modified radical mastectomy. Patients with close margins (tumor < 1 mm from margin) are eligible.
     * Segmental mastectomy (lumpectomy): Although clear margins are preferable, DCIS or LCIS at the surgical resection margin will not render a patient who has undergone a segmental mastectomy ineligible for this study. Invasive tumor at the final resection margin will render a patient ineligible.
   * No prior chemotherapy for this malignancy.
   * Patients with a history of hypersensitivity to 5-FU or known dihydropyrimidine dehydrogenase (DPD) deficiency are not eligible to participate.
   * Patients may receive up to four weeks of tamoxifen therapy for this malignancy and still be eligible for study entry. Patients who received tamoxifen or raloxifene for purposes of chemoprevention (e.g., Breast Cancer Prevention Trial) or for other indications (including previous breast cancer) are eligible. Tamoxifen or raloxifene therapy should be discontinued before the patient is enrolled on this study.
7. Required Initial Laboratory Data:

   * Granulocytes > 1,500/µl
   * Platelet count ≥100,000/µl
   * Calculated Creatinine Clearance > 30 mL/min
   * Total bilirubin ≤ ULN

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 633 (Actual)
Dates: Start 2001-09; Primary Completion 2008-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyman B. Muss, MD, Study Chair — University of North Carolina
Locations (334):
- United States (326):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - St. Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Saint Rose Hospital, Hayward, California
  - Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Kent General Hospital at Bayhealth Medical Center, Dover, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Halifax Medical Center - Daytona Beach, Daytona Beach, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Palm Beach Cancer Institute - West Palm Beach, West Palm Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Maui, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Wasser Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Regional Cancer Institute at Bloomington Hospital, Bloomington, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Community Hospital, Munster, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology & Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Mercy Hospital of Portland, Portland, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - MaineGeneral Medical Center - Waterville Campus, Waterville, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Saints Memorial Cancer Center at Saints Memorial Medical Center, Lowell, Massachusetts
  - Lawrence Memorial Hospital of Medford, Medford, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Carson-Tahoe Cancer Services at Carson Tahoe Regional Healthcare, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Parkland Oncology-Hematology Clinic at Parkland Medical Center, Derry, New Hampshire
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Winthrop University Hospital, Mineola, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Bronx-Lebanon Hospital Center & BronxCare Adult Medical Practice, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Nashville Oncology Associates, P.C., Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Marshall University Medical Center, Huntington, West Virginia
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (7):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Prince Edward Island Cancer Centre at Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- [Background] Pal SK, Mortimer J. Adjuvant chemotherapy for older adults with breast cancer: making the standard a standard. Womens Health (Lond). 2009 Sep;5(5):481-4. doi: 10.2217/whe.09.43. PMID 19702447
- [Result] Partridge AH, Archer L, Kornblith AB, Gralow J, Grenier D, Perez E, Wolff AC, Wang X, Kastrissios H, Berry D, Hudis C, Winer E, Muss H. Adherence and persistence with oral adjuvant chemotherapy in older women with early-stage breast cancer in CALGB 49907: adherence companion study 60104. J Clin Oncol. 2010 May 10;28(14):2418-22. doi: 10.1200/JCO.2009.26.4671. Epub 2010 Apr 5. PMID 20368559
- [Result] Kornblith AB, Archer L, Lan L, et al.: Quality of life of early stage breast cancer patients 65 years old or older randomized to standard chemotherapy or capecitabine: A Cancer and Leukemia Group B Study (CALGB 49907). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-5035, 2009.
- [Result] Muss HB, Berry DA, Cirrincione CT, Theodoulou M, Mauer AM, Kornblith AB, Partridge AH, Dressler LG, Cohen HJ, Becker HP, Kartcheske PA, Wheeler JD, Perez EA, Wolff AC, Gralow JR, Burstein HJ, Mahmood AA, Magrinat G, Parker BA, Hart RD, Grenier D, Norton L, Hudis CA, Winer EP; CALGB Investigators. Adjuvant chemotherapy in older women with early-stage breast cancer. N Engl J Med. 2009 May 14;360(20):2055-65. doi: 10.1056/NEJMoa0810266. PMID 19439741
- [Result] Muss HB, Berry DL, Cirrincione C, et al.: Standard chemotherapy (CMF or AC) versus capecitabine in early-stage breast cancer (BC) patients aged 65 and older: results of CALGB/CTSU 49907. [Abstract] J Clin Oncol 26 (Suppl 15): A-507, 2008.
- [Result] Partridge AH, Archer LE, Kornblith AB, et al.: CALGB 60104: adherence with adjuvant capecitabine among women age 65 and older with early stage breast cancer treated on CALGB 49907. [Abstract] J Clin Oncol 26 (Suppl 15): A-6542, 2008.
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Muss HB, Polley MC, Berry DA, Liu H, Cirrincione CT, Theodoulou M, Mauer AM, Kornblith AB, Partridge AH, Dressler LG, Cohen HJ, Kartcheske PA, Perez EA, Wolff AC, Gralow JR, Burstein HJ, Mahmood AA, Sutton LM, Magrinat G, Parker BA, Hart RD, Grenier D, Hurria A, Jatoi A, Norton L, Hudis CA, Winer EP, Carey L. Randomized Trial of Standard Adjuvant Chemotherapy Regimens Versus Capecitabine in Older Women With Early Breast Cancer: 10-Year Update of the CALGB 49907 Trial. J Clin Oncol. 2019 Sep 10;37(26):2338-2348. doi: 10.1200/JCO.19.00647. Epub 2019 Jul 24. PMID 31339827
- [Derived] Magnuson A, Lei L, Gilmore N, Kleckner AS, Lin FV, Ferguson R, Hurria A, Wittink MN, Esparaz BT, Giguere JK, Misleh J, Bautista J, Mohile SG, Janelsins MC. Longitudinal Relationship Between Frailty and Cognition in Patients 50 Years and Older with Breast Cancer. J Am Geriatr Soc. 2019 May;67(5):928-936. doi: 10.1111/jgs.15934. PMID 31034595
- [Derived] Gajra A, McCall L, Muss HB, Cohen HJ, Jatoi A, Ballman KV, Partridge AH, Sutton L, Parker BA, Magrinat G, Klepin HD, Lafky JM, Hurria A. The preference to receive chemotherapy and cancer-related outcomes in older adults with breast cancer CALGB 49907 (Alliance). J Geriatr Oncol. 2018 May;9(3):221-227. doi: 10.1016/j.jgo.2018.02.003. Epub 2018 Mar 28. PMID 29602735
- [Derived] Morrison VA, McCall L, Muss HB, Jatoi A, Cohen HJ, Cirrincione CT, Ligibel JA, Lafky JM, Hurria A. The impact of actual body weight-based chemotherapy dosing and body size on adverse events and outcome in older patients with breast cancer: Results from Cancer and Leukemia Group B (CALGB) trial 49907 (Alliance A151436). J Geriatr Oncol. 2018 May;9(3):228-234. doi: 10.1016/j.jgo.2017.11.007. Epub 2017 Dec 8. PMID 29233548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an intergroup study led by the CALGB. Between September 2001 and December 2006, 633 participants were recruited.
Pre-assignment Details: All participants recruited were randomized with equal probability to one of two treatment arms. Randomization was initially stratified by age and performance score. In 2006 tumoral HER2 status was added as a third stratification factor.
Groups:
- Standard Chemotherapy: Patient/Physician choice of:
  CMF: cyclophosphamide (100 mg/m^2 orally days 1-14)+ MTX (40 mg/m^2 by IV days 1 and 8) + 5-FU (600 mg/m^2 by IV days 1 and 8) repeated every 28 days for 6 cycles
  OR
  AC: Cyclophosphamide (600 mg/m^2 by IV on day 1)+ doxorubicin (60 mg/m^2 by IV on day 1) repeated every 21 days for 4 cycles
- Capecitabine: Capecitabine (2000 mg/m^2 in 2 doses days 1-14) repeated every 21 days for 6 cycles.
Period: Overall Study
Arm/Group | Standard Chemotherapy | Capecitabine
Started | 326 | 307
Completed | 326 | 307
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Chemotherapy | Capecitabine | Total
Number analyzed (Participants) | 326 | 307 | 633
Age, Customized [Number; unit: participants]
  65-69 years | 112 | 110 | 222
  70-79 years | 200 | 183 | 383
  >=80 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 307 | 633
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 326 | 302 | 628
  Argentina | 0 | 3 | 3
  Australia | 0 | 2 | 2
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 or 1 (fully active or minimal symptoms) | 317 | 295 | 612
    2 (symptoms, but active > 50% of the time) | 9 | 12 | 21
HER2 Status [Number; unit: participants]
  Negative | 246 | 232 | 478
  Positive | 35 | 30 | 65
  Unknown | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival Rates at 2.4 Years
Description: Percentage of participants who were alive and relapse-free at time of analysis were counted as "Alive without relapse" at 2.4 years. Participants who had a first local recurrence, first distant metastasis or death from any cause were counted as "relapse, first occurrence". These rates were estimated using the Kaplan Meier method
Time Frame: randomization until date of first event, or date last known to be event free if no event was reported (up to 5 years)
Population: RFS used the intent-to-treat approach
Measure: Number; unit: percentage of participants
Arm/Group | Standard Chemotherapy | Capecitabine
Number analyzed (Participants) | 326 | 307
percentage of participants
  Relapse, first occurrence | 11 | 20
  Alive without relapse | 89 | 80
Statistical Analysis 1: Comparison: Standard Chemotherapy vs Capecitabine; Test type: Non-Inferiority or Equivalence — The primary measure of efficacy was the hazard ratio for disease recurrence or death in the capecitabine group as compared with the standard chemotherapy group. Capecitabine would be considered noninferior to standard chemotherapy if the hazard ratio was greater than 0.8046. (With the use of a 5-year landmark for descriptive purposes, this ratio corresponds to a 5-year rate of relapse-free survival of 60% for standard chemotherapy and 53% for capecitabine.); p < 0.001, Regression, Cox — Multivariate proportional hazards regression used to test for an arm effect was adjusted for tumor size, number of lymph nodes and hormone-receptor status. A priori formal monitoring for futility and noninferiority was planned at accrual milestones; Hazard Ratio (HR) = 2.09, 95% CI 2-sided [1.38 to 3.17]

2. Secondary Outcome: Overall Survival Rate at 2.4 Years
Description: Percentage of patients who were alive at 2.4 years. This rate was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death (up to 15 years)
Population: OS used the intent-to-treat approach.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Chemotherapy | Capecitabine
Number analyzed (Participants) | 326 | 307
percentage of participants | 93 | 88
Statistical Analysis 1: Comparison: Standard Chemotherapy vs Capecitabine; Test type: Superiority or Other; p = 0.02, Regression, Cox — Multivariate proportional hazards regression used to test for an arm effect was adjusted for tumor size, number of lymph nodes and hormone-receptor status. There is no adjustment for multiple comparisons; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [1.11 to 3.08]

3. Secondary Outcome: Number of Participants With Grade 3, 4 or 5 Adverse Event at Least Possibly Related to Treatment.
Description: The National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Version 2.0 was used to evaluate toxicity.
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: Reported during protocol treatment after each cycle
Measure: Number; unit: participants
Groups:
- Standard Chemotherapy (CMF): CMF: cyclophosphamide (100 mg/m^2 orally days 1-14)+ MTX (40 mg/m^2 by IV days 1 and 8) + 5-FU (600 mg/m^2 by IV days 1 and 8) repeated every 28 days for 6 cycles
- Standard Chemotherapy (AC): AC: Cyclophosphamide (600 mg/m^2 by IV on day 1)+ doxorubicin (60 mg/m^2 by IV on day 1) repeated every 21 days for 4 cycles
Arm/Group | Standard Chemotherapy (CMF) | Standard Chemotherapy (AC) | Capecitabine
Number analyzed (Participants) | 132 | 183 | 299
participants | 92 | 109 | 101

ADVERSE EVENTS:
Time Frame: Reported at the end of each cycle while patients were receiving protocol therapy.
Arm/Group | Standard Chemotherapy (CMF) | Standard Chemotherapy (AC) | Capecitabine
Serious Adverse Events (participants affected / at risk) | 15/131 | 17/181 | 26/299
Other Adverse Events (participants affected / at risk) | 121/131 | 168/181 | 279/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemotherapy (CMF) (N=131) | Standard Chemotherapy (AC) (N=181) | Capecitabine (N=299)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (7) | 13 (13) | 8 (9)
Lymphatics (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 5 (5) | 18 (20)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 10 (10)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (8) | 9 (9) | 16 (20)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 4 (4)
INR increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 12 (13) | 13 (14) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (8) | 10 (11) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 8 (8) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 10 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 7 (7)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rash/Dermatitis BMT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (11)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Peripheral arterial ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemotherapy (CMF) (N=131) | Standard Chemotherapy (AC) (N=181) | Capecitabine (N=299)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 18 (22) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 54 (158) | 112 (293) | 67 (199)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphatics (Blood and lymphatic system disorders) | 17 (35) | 4 (5) | 23 (44)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 1 (1) | 7 (9)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 2 (4)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Flashing vision (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (10)
Diarrhea (Gastrointestinal disorders) | 58 (108) | 32 (52) | 138 (276)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 38 (61) | 58 (89) | 71 (117)
Nausea (Gastrointestinal disorders) | 66 (151) | 105 (201) | 102 (185)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (40) | 40 (48) | 29 (34)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 86 (299) | 129 (321) | 162 (504)
Fever (General disorders) | 2 (2) | 2 (2) | 0 (0)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (5) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 5 (5) | 1 (2)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Infection without neutropenia (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (4)
Alanine aminotransferase increased (Investigations) | 3 (7) | 0 (0) | 5 (6)
Alkaline phosphatase (Investigations) | 1 (3) | 0 (0) | 2 (6)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 0 (0) | 5 (9)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 3 (4)
Creatinine increased (Investigations) | 10 (14) | 6 (10) | 22 (46)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 4 (6) | 0 (0) | 3 (11)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 87 (256) | 112 (270) | 31 (71)
Lymphocyte count decreased (Investigations) | 6 (9) | 4 (8) | 1 (1)
Neutrophil count decreased (Investigations) | 37 (66) | 54 (106) | 5 (8)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Investigations) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 46 (105) | 47 (83) | 11 (13)
Platelets for BMT studies, if specified in the protocol. (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (4) | 3 (5) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 36 (64) | 41 (67) | 52 (92)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (25) | 10 (16) | 12 (23)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (6) | 3 (4) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (4) | 1 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 3 (5) | 6 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (6)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 4 (8) | 0 (0) | 3 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (2) | 4 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 5 (9)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 0 (0) | 6 (10)
Sense of smell (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (3) | 4 (5) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (7) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5) | 4 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (10) | 5 (6) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 8 (15) | 2 (2) | 210 (657)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 13 (20) | 15 (25) | 55 (109)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 4 (6)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 5 (5) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes